CLINICAL TRIAL: NCT03930979
Title: The Effect of Hyperoxia on Cardiac Output in Patients Undergoing Procedural Sedation in the Emergency Department.
Brief Title: The Effect of Hyperoxia on Cardiac Output
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: nWMO270
Record Dates: First submitted 2018-07-17; First posted 2019-04-29 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2019-08

CONDITIONS: Hyperoxia; Cardiac Output, Low
Keywords: Procedural sedation; Cardiac output measurements non-invasive; Emergency department
MeSH Terms: conditions — Hyperoxia; Cardiac Output, Low; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clearsight measurements: All patients presenting to the ED who have a painful condition for which procedural sedation is required will undergo Clearsight measurements

SUMMARY:
Rational: Preoxygenation is a standard procedure before (deep) sedation in the ED. However, there is literature suggesting that too much oxygen can be harmful. One potential detrimental effect is a decrease in cardiac output due to coronary vasoconstriction. So far, it is unknown if this effect is rate dependent and if it also occurs after only a short period of hyperoxia, as patients experience during procedural sedation pre-oxygenation.

Objective: To investigate if hyperoxia has a negative effect on Cardiac index (CI) in patients undergoing procedural sedation in the ED.

DETAILED DESCRIPTION:
Methods: In patients needing sedation for a painful condition, non-invasive measurements of CI, stroke volume and total peripheral resistance are performed using the Clearsight non-invasive cardiac output monitoring system.. Measurements will be taken at baseline, after 1,2 and 5 minutes of 15L O2/min, and then after another 2 and 5 minutes of flush rate oxygen and during the subsequent sedation.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting in the ED of the Medical Center Leeuwarden (MCL) who have a painful condition for which procedural sedation is required.

Exclusion Criteria:

* - Cardiogenic shock (SBP<90 mmHg)
* Procedural sedation for cardioversion
* Pregnancy
* General contra-indications for the procedural sedation according to local sedation protocol of the MCL.
* Hypoxia (sat <90% or pO2 <8)) despite oxygen suppletion
* Age < 18 years
* Non-invasive ventilation (NIV) or intubation
* No informed consent
* Use of bleomycin
* COPD GOLD III of IV
* COPD GOLD I of II with hypercapnia (PCO2 > 6,4 kPa)
* Patients in whom no reliable signal for Clearsight measurement can be obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patients presenting in the ED of the Medical Center Leeuwarden (MCL) who have a painful condition for which procedural sedation is required.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
The change in cardiac output (L/min) after respectively 15L/min and flush rate preoxygenation in respect to baseline | at baseline, at 1,2,5 (15L),7 and 10 minutes (flush o2)
  Cardiac output is measured by Clearsight non invasive hemodynamic monitoring system; 3 baseline measurements are done separated by one minute intervals; subsequently 15L/min O2 is started. After 1,2 and 5 minutes, measurements are repeated. After 5 minutes, flush rate O2 is started. After 2 and 5 minutes, measurements are repeated.

SECONDARY OUTCOMES:
The change in heart rate (BPM) after respectively 15L/min and flush rate preoxygenation in respect to baseline | at baseline, at 1,2,5, (15L o2) and 7, 10 minutes (flush o2)
  3 baseline measurements are done separated by one minute intervals; subsequently 15L/min O2 is started. After 1,2 and 5 minutes, measurements are repeated. After 5 minutes, flush rate O2 is started. After 2 and 5 minutes, measurements are repeated.
the change in systolic blood pressure (mmHg) after respectively 15L/min and flush rate preoxygenation in respect to baseline | at baseline, at 1,2,5 (15L o2) and 7, 10 minutes (flush o2)
  Systolic blood pressure is measured by Clearsight non invasive hemodynamic monitoring system; 3 baseline measurements are done separated by one minute intervals; subsequently 15L/min O2 is started. After 1,2 and 5 minutes, measurements are repeated. After 5 minutes, flush rate O2 is started. After 2 and 5 minutes, measurements are repeated.
The change in stroke volume (ml) after respectively 15L/min and flush rate preoxygenation in respect to baseline | at baseline, at 1,2,5 (15L o2) and 7, 10 minutes (flush o2)
  Stroke volume is measured by Clearsight non invasive hemodynamic monitoring system; 3 baseline measurements are done separated by one minute intervals; subsequently 15L/min O2 is started. After 1,2 and 5 minutes, measurements are repeated. After 5 minutes, flush rate O2 is started. After 2 and 5 minutes, measurements are repeated.
the change in total peripheral vascular resistance after respectively 15L/min and flush rate preoxygenation in respect to baseline | at baseline, at 1,2,5 (15L o2) and 7,10 minutes (flush o2)
  Peripheral vascular resistance is measured by Clearsight non invasive hemodynamic monitoring system; 3 baseline measurements are done separated by one minute intervals; subsequently 15L/min O2 is started. After 1,2 and 5 minutes, measurements are repeated. After 5 minutes, flush rate O2 is started. After 2 and 5 minutes, measurements are repeated.
The relation of the difference in CI with the occurrence of of haemodynamic sedation events | at baseline, at 1,2,5 (15L o2) ,7 and 10 minutes (flush o2)
  In case of apnea > 20 sec, low SBP <90 mmHg or >20% decrease in comparison to baseline, desaturation <92%, assess relation to change in cardiac output (L/min) during preoxygenation

CONTACTS AND LOCATIONS:
Overall Officials: Ewoud ter Avest, MD, PhD, Principal Investigator — medical center leeuwarden; Renate Stolmeijer, MD, Principal Investigator — medical center leeuwarden
Locations (1):
- Medical Center Leeuwarden, Leeuwarden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided